CLINICAL TRIAL: NCT04548947
Title: Does Routine Submucosal Injection Improve Complete Resection of 4-20 mm Neoplastic Colorectal Polyps?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20.111
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; incomplete resection rate; submucosal injection; neoplastic polyps
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: prospective, multi-endoscopist, single center, clinical study at tertiary referral center (CHUM)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cold snare polypectomy with a submucosal injection (Experimental): The procedure will include a cold snare polypectomy with a submucosal injection done prior to the resection.
  Interventions: Procedure: Cold snare polypectomy in conjunction with a submucosal injection

INTERVENTIONS:
Procedure: Cold snare polypectomy in conjunction with a submucosal injection — The cold snare polypectomy in conjunction with a submucosal injection is a procedure during which the endoscopist resects the colorectal polyps during a colonoscopy, without any electrocautery.

SUMMARY:
This is a prospective, multi-endoscopist, single center, clinical study at tertiary referral center that addresses an important current challenge in the prevention of colorectal cancer (CRC), namely, how to improve the complete removal of CRC precursors. This study will observe the potential benefit of specific polypectomy technique in conjunction with a systematic submucosal injection prior to the polyp resection. This study will evaluate the completeness and incompleteness of the resection of colorectal neoplastic polyps during the procedures.

DETAILED DESCRIPTION:
Non-detection and incomplete resection of neoplastic colorectal polyps have been identified as the main risk factors for the development of CRC in patients after a colonoscopy. Between 7% and 9% of all newly diagnosed CRCs are estimated to be such "interval cancers," occurring after a previous colonoscopy and before the next surveillance examination. The vast majority of interval cancers are caused by incomplete detection or resection during colonoscopy examination. The contribution of incomplete resection towards interval cancer has recently been pointed out by a panel of experts as one of the cornerstones of CRC prevention that need to be addressed in future research studies. The primary aim of this study is to examine the incomplete adenoma resection rates when performing a cold snare polypectomy in conjunction with a submucosal injection for endoscopic resection of 4-20 mm non-pedunculated colorectal polyps. The subjects are patients, men and women, aged between 45-80 years old that are scheduled for a colonoscopy. The secondary aims are to identify procedure-related complication rates and patient-, polyp-, and endoscopist-related factors associated with incomplete adenoma resection.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form; aged 45-80 years old, indication to undergo a colonoscopy

Exclusion Criteria:

* Known inflammatory bowel disease; active colitis; coagulopathy; familial polyposis syndrome; poor general health, defined as an American Society of Anesthesiologists (ASA) physical status class >3; emergency colonoscopies, hospitalized patients or patients referred from the emergency room.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Incomplete resection rate (IRR) | Day 1
  The number of incomplete polyps resected after polypectomy, as defined by any neoplastic tissue found in marginal biopsies.

SECONDARY OUTCOMES:
Immediate bleeding complications | Day 1
  bleeding requiring endoscopic intervention either during colonoscopy/polypectomy, or requiring an immediate second intervention such as surgery and/or hospital admission
Delayed bleeding complications | 14 days after the initial procedure
  bleeding after the end of the initial procedure 14 days later
Other severe complications | 14 days after the initial procedure
  Post-polypectomy syndrome and perforation requiring endoscopic intervention and/or surgery, and/or hospital admission
Proportion of polyps considered interpretable for complete polyp removal | 14 days after the initial procedure
  Proportion of polyps considered interpretable for complete polyp removal
Incomplete resection of colorectal polyps | 14 days after the initial procedure
  Incomplete resection rates of colorectal polyps after widefield resection (defined as resection margins of the largest of 3mm or 25% of the resected polyp size) of 1-20mm polyps using SCALE-EYE as measurement tool vs standard non wide field polypectomy (defined by positive tissue remnants at biopsy sites [vertical and lateral margins, 4 biopsies])

CONTACTS AND LOCATIONS:
Overall Officials: Daniel von Renteln, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier Universitaire de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No